CLINICAL TRIAL: NCT05896501
Title: Role of Fractional Flow Reserve Assessment Using Pressure Wire in Patients With Acute Coronary Syndrome Who Treated With Xience Stent; a Multicenter, Prospective, and Observational Registry
Brief Title: Role of FFR in ACS Patients: Pressure ACS Registry
Status: Active, not recruiting | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Eun Ho Choo, Assistant Professor, The Catholic University of Korea
Other Study IDs: PressureACS
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fractional Flow Reserve — Functional assessement of anatomical stenosis of coronary artery

SUMMARY:
Currently, fractional flow reserve (FFR) is regarded as a gold-standard invasive method to define lesion-specific ischemia and FFR-guided PCI has been proven to reduce unnecessary revascularization and to enhance patient's clinical outcomes. Therefore, current guidelines recommend FFR measurement for intermediate coronary stenosis when there is no definite evidence of lesion-specific ischemia. However, previous evidences which well demonstrated the benefit of FFR-guided strategy were mostly generated from patients with stable coronary artery disease.4 FFR may be overestimated and the hemodynamic relevance of a coronary stenosis underestimated in patients with acute coronary syndrome (ACS).Its role in ACS patients still needs to be defined although several studies have recently published addressing the value of FFR-guided PCI in ACS. In fact, recent evidence suggests that culprit lesions of patients presenting with a non-ST-segment elevation myocardial infarction that were deferred based on a "negative" FFR have a relatively high event rate, calling into question the use of FFR in that patient population.

DETAILED DESCRIPTION:
STUDY OBJECTIVE

1. To evaluate the impact of FFR on decision for PCI in ACS patients
2. To assess the long term prognosis of deferring PCI based on FFR value in non-culprit lesion; defying the cut-off value of FFR for PCI in the non-culprit lesion of ACS patients
3. To identify the relation between OCT findings and FFR value in culprit and non-culprit lesions of ACS patients
4. To compare the long term prognosis of PCI or deferring PCI based on FFR value in non-culprit lesion of ACS patients
5. To identify OCT findings to predict the lesion progression in deferred lesions.
6. To assess the long term prognosis of post-PCI FFR value in the culprit lesion of NSTE-ACS patients
7. To assess the efficacy of routine use of FFR to guide PCI in ACS patients; angiographically guidance versus FFR guidance

ELIGIBILITY:
Inclusion Criteria:

* Subject age 19-85 years old

  * Diagnosed as ACS (unstable angina/ Non ST elevation myocardial infarction, ST elevation myocardial infarction)

    * At least one stenosis of >50% in a non-culprit vessel ≥ 2.0 mm by visual estimation with TIMI 3 - multivessel disease after PCI for culprit lesion or single vessel disease with ambiguity for PCI ④ FFR within hospitalization for index PCI for ACS

Exclusion Criteria:

* Severe stenosis with TIMI flow ≤ II of the non-IRA artery

  * Cardiogenic shock (Killip class IV) already at presentation or the completion of culprit PCI

    * Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparin, Bivaluridin, or Everolimus

      * Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)

        ⑤ Pregnancy or breast feeding

        ⑥ Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol noncompliance (per site investigator's medical judgment).

        ⑦ Other primary valvular disease with severe degree: severe mitral regurgitation or mitral stenosis, severe aortic regurgitation or aortic stenosis

        ⑧ Patients with a history of Coronary Artery Bypass Graft(CABG)

        ⑨ Unwillingness or inability to comply with the procedures described in this protocol.

Ages: 19 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome and intermediate stenosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Major adverse cardiac events | 24 months
  Rate of the composite of all-cause death, recurrent myocardial infarction

SECONDARY OUTCOMES:
Rate of Major adverse cardiac events at 1 year | 12 months
  Rate of composite of all-cause death, recurrent myocardial infarction
Rate of Ischemic events | 24 months
  Rate of the composite of all-cause death, recurrent myocardial infarction, and any repeat revascularization
Rate of Death | 24 months
  Rate of All cause death and cardiac death
Rate of Repeat revascularization | 24 months
  Rate of Any repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Eun Ho Choo, M.D.,PhD, Principal Investigator — The Catholic University of Korea
Locations (5):
- South Korea (5):
  - St.Vincent's Hospital, Suwon, Gyeonggido
  - Uijeongbu St.Mary's Hospital, Uijeongbu-si, Gyeonggido
  - Daejeon St.Mary's Hospital, Daejeon
  - Incheon St.Mary's Hospital, Incheon
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided